CLINICAL TRIAL: NCT00262522
Title: A Phase 3, Randomized, Open-label, Study of Lopinavir/Ritonavir Tablets Versus Soft Gel Capsules and Once Daily Versus Twice Daily Administration, When Coadministered With NRTIs in Antiretroviral Naive HIV-1 Infected Subjects
Brief Title: Study of Lopinavir/Ritonavir Tablets Versus Soft Gel Capsules and Once Daily Versus Twice Daily Administration, When Coadministered With Nucleoside Reverse Transcriptase Inhibitors in Antiretroviral Naive Human Immunodeficiency Virus Type 1 Infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M05-730; 2005-001430-32 (EudraCT Number)
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Results first posted 2009-08-20 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Human Immunodeficiency Virus Infections
Keywords: Human Immunodeficiency Virus Infections
MeSH Terms: interventions — Lopinavir; Ritonavir; Tablets; Capsules; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LPV/r 800/200 mg QD Tablet (Experimental)
  Interventions: Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs)
- LPV/r 800/200 mg QD SGC (Through Week 8) (Experimental)
  Interventions: Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs)
- LPV/r 400/100 mg BID Tablet (Active Comparator)
  Interventions: Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs)
- LPV/r 400/100 mg BID SGC (Through Week 8) (Active Comparator)
  Interventions: Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs)

INTERVENTIONS:
Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs) — LPV/r 800/200 mg once daily (QD) tablet + emtricitabine (FTC) 200 mg QD + tenofovir disoproxil fumarate (TDF) 300 mg QD
  Other Names: ABT-378, Kaletra, lopinavir/ritonavir
  Arms: LPV/r 800/200 mg QD Tablet
Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs) — LPV/r 800/200 mg QD soft gel capsule (SGC) + FTC 200 mg QD + TDF 300 mg QD (8 weeks) followed by LPV/r 800/200 mg QD Tablet + FTC 200 mg QD + TDF 300 mg QD
  Other Names: ABT-378, Kaletra, lopinavir/ritonavir
  Arms: LPV/r 800/200 mg QD SGC (Through Week 8)
Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs) — LPV/r 400/100 mg twice daily (BID) tablet + FTC 200 mg QD + TDF 300 mg QD
  Other Names: ABT-378, Kaletra, lopinavir/ritonavir
  Arms: LPV/r 400/100 mg BID Tablet
Drug: lopinavir/ritonavir (LPV/r) (tablet or capsule) with nucleoside reverse transcriptase inhibitors (NRTIs) — LPV/r 400/100 mg BID SGC + FTC 200 mg QD + TDF 300 mg QD (8 weeks) followed by LPV/r 400/100 mg BID Tablet + FTC 200 mg QD + TDF 300 mg QD
  Other Names: ABT-378, Kaletra, lopinavir/ritonavir
  Arms: LPV/r 400/100 mg BID SGC (Through Week 8)

SUMMARY:
The purpose of this study was to compare the safety and tolerability of the to-be-marketed lopinavir/ritonavir (LPV/r) tablet formulation with the marketed soft gel capsule (SGC) formulation and to compare the safety, tolerability, and antiviral activity of once daily (QD) and twice daily (BID) dosing of the LPV/r tablet formulation in combination with select nucleoside reverse transcriptase inhibitors (NRTIs) in patients who have not previously received antiretroviral treatment.

ELIGIBILITY:
Inclusion Criteria

* Subjects were human immunodeficiency virus type 1 (HIV-1) positive, antiretroviral naïve adults at least 18 years of age with < 7 days of prior antiretroviral therapy.
* Subjects had plasma HIV-1 ribonucleic acid (RNA) levels >= 1,000 copies/mL at screening and were not acutely ill.
* Female subjects were nonpregnant and nonlactating.

Exclusion Criteria

* Subjects were excluded if screening laboratory analyses showed any of the following abnormal laboratory results:

  * Presence of hepatitis B surface antigen (HBsAg)
  * Hemoglobin <= 8.0 g/dL
  * Absolute neutrophil count <= 750 cells/microliter
  * Platelet count <= 50,000 per mL
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >= 3.0 x Upper Limit of Normal (ULN)
  * Calculated creatinine clearance < 50 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Cohen, MD, Study Director — Abbott
Locations (129):
- United States (30):
  - Site Reference ID/Investigator# 823, Phoenix, Arizona
  - Site Reference ID/Investigator# 846, Phoenix, Arizona
  - Site Reference ID/Investigator# 851, Beverly Hills, California
  - Site Reference ID/Investigator# 872, Fountain Valley, California
  - Site Reference ID/Investigator# 826, Long Beach, California
  - Site Reference ID/Investigator# 876, Newport Beach, California
  - Site Reference ID/Investigator# 875, Washington D.C., District of Columbia
  - Site Reference ID/Investigator# 870, Atlantis, Florida
  - Site Reference ID/Investigator# 844, Fort Lauderdale, Florida
  - Site Reference ID/Investigator# 874, Miami, Florida
  - Site Reference ID/Investigator# 1153, Orlando, Florida
  - Site Reference ID/Investigator# 827, Orlando, Florida
  - Site Reference ID/Investigator# 783, Plantation, Florida
  - Site Reference ID/Investigator# 877, Port Saint Lucie, Florida
  - Site Reference ID/Investigator# 845, Safety Harbor, Florida
  - Site Reference ID/Investigator# 849, Sarasota, Florida
  - Site Reference ID/Investigator# 825, Tampa, Florida
  - Site Reference ID/Investigator# 848, Atlanta, Georgia
  - Site Reference ID/Investigator# 873, Macon, Georgia
  - Site Reference ID/Investigator# 1154, Chicago, Illinois
  - Site Reference ID/Investigator# 824, Chicago, Illinois
  - Site Reference ID/Investigator# 792, Wichita, Kansas
  - Site Reference ID/Investigator# 1157, Minneapolis, Minnesota
  - Site Reference ID/Investigator# 871, St Louis, Missouri
  - Site Reference ID/Investigator# 2450, Rochester, New York
  - Site Reference ID/Investigator# 784, Charlotte, North Carolina
  - Site Reference ID/Investigator# 1155, Dallas, Texas
  - Site Reference ID/Investigator# 850, Dallas, Texas
  - Site Reference ID/Investigator# 843, Houston, Texas
  - Site Reference ID/Investigator# 1156, Hampton, Virginia
- Australia (3):
  - Site Reference ID/Investigator# 244, Darlinghurst
  - Site Reference ID/Investigator# 245, Melbourne
  - Site Reference ID/Investigator# 246, South Yarra
- Belgium (5):
  - Site Reference ID/Investigator# 234, Antwerp
  - Site Reference ID/Investigator# 235, Brussels
  - Site Reference ID/Investigator# 233, Ghent
  - Site Reference ID/Investigator# 236, Leuven
  - Site Reference ID/Investigator# 225, Liège
- Canada (13):
  - Site Reference ID/Investigator# 175, Calgary
  - Site Reference ID/Investigator# 184, Hamilton
  - Site Reference ID/Investigator# 177, Montreal
  - Site Reference ID/Investigator# 176, Montreal
  - Site Reference ID/Investigator# 179, Montreal
  - Site Reference ID/Investigator# 181, Ottawa
  - Site Reference ID/Investigator# 173, Ottawa
  - Site Reference ID/Investigator# 178, Ste-Foy
  - Site Reference ID/Investigator# 180, Toronto
  - Site Reference ID/Investigator# 182, Toronto
  - Site Reference ID/Investigator# 174, Toronto
  - Site Reference ID/Investigator# 183, Vancouver
  - Site Reference ID/Investigator# 172, Vancouver
- Czechia (2):
  - Site Reference ID/Investigator# 294, Brno
  - Site Reference ID/Investigator# 296, Pilsen
- France (11):
  - Site Reference ID/Investigator# 286, Aix-en-Provence
  - Site Reference ID/Investigator# 275, Besançon
  - Site Reference ID/Investigator# 256, Lyon
  - Site Reference ID/Investigator# 278, Montpellier
  - Site Reference ID/Investigator# 257, Paris
  - Site Reference ID/Investigator# 281, Paris
  - Site Reference ID/Investigator# 280, Paris
  - Site Reference ID/Investigator# 279, Paris
  - Site Reference ID/Investigator# 284, Paris
  - Site Reference ID/Investigator# 274, Rennes
  - Site Reference ID/Investigator# 282, Vandœuvre-lès-Nancy
- Germany (10):
  - Site Reference ID/Investigator# 265, Berlin
  - Site Reference ID/Investigator# 270, Berlin
  - Site Reference ID/Investigator# 262, Bochum
  - Site Reference ID/Investigator# 268, Bonn
  - Site Reference ID/Investigator# 271, Cologne
  - Site Reference ID/Investigator# 266, Frankfurt
  - Site Reference ID/Investigator# 264, Fürth
  - Site Reference ID/Investigator# 273, Hamburg
  - Site Reference ID/Investigator# 267, Hamburg
  - Site Reference ID/Investigator# 263, Hanover
- Greece (2):
  - Site Reference ID/Investigator# 211, Athens
  - Site Reference ID/Investigator# 207, Thessaloniki
- Ireland (2):
  - Site Reference ID/Investigator# 237, Dublin
  - Site Reference ID/Investigator# 249, Dublin
- Italy (10):
  - Site Reference ID/Investigator# 203, Brescia
  - Site Reference ID/Investigator# 192, Florence
  - Site Reference ID/Investigator# 195, Genoa
  - Site Reference ID/Investigator# 201, Milan
  - Site Reference ID/Investigator# 198, Milan
  - Site Reference ID/Investigator# 199, Pavia
  - Site Reference ID/Investigator# 200, Rome
  - Site Reference ID/Investigator# 196, Rome
  - Site Reference ID/Investigator# 194, Rome
  - Site Reference ID/Investigator# 193, Turin
- Site Reference ID/Investigator# 290, Zwolle, Netherlands
- Poland (3):
  - Site Reference ID/Investigator# 298, Chorzów
  - Site Reference ID/Investigator# 299, Warsaw
  - Site Reference ID/Investigator# 297, Wroclaw
- Puerto Rico (3):
  - Site Reference ID/Investigator# 185, Ponce
  - Site Reference ID/Investigator# 208, Ponce
  - Site Reference ID/Investigator# 206, San Juan
- Russia (3):
  - Site Reference ID/Investigator# 186, Moscow
  - Site Reference ID/Investigator# 189, Moscow
  - Site Reference ID/Investigator# 188, Saint Petersburg
- Site Reference ID/Investigator# 5163, Singapore, Singapore
- Spain (18):
  - Site Reference ID/Investigator# 221, A Coruña
  - Site Reference ID/Investigator# 210, Alicante
  - Site Reference ID/Investigator# 190, Barakaldo
  - Site Reference ID/Investigator# 214, Barcelona
  - Site Reference ID/Investigator# 216, Barcelona
  - Site Reference ID/Investigator# 222, Barcelona
  - Site Reference ID/Investigator# 224, Barcelona
  - Site Reference ID/Investigator# 218, Barcelona
  - Site Reference ID/Investigator# 292, Madrid
  - Site Reference ID/Investigator# 205, Madrid
  - Site Reference ID/Investigator# 191, Madrid
  - Site Reference ID/Investigator# 219, Madrid
  - Site Reference ID/Investigator# 209, Madrid
  - Site Reference ID/Investigator# 223, Madrid
  - Site Reference ID/Investigator# 213, Santander
  - Site Reference ID/Investigator# 217, Santiago de Compostela
  - Site Reference ID/Investigator# 220, Seville
  - Site Reference ID/Investigator# 215, Valencia
- Switzerland (4):
  - Site Reference ID/Investigator# 288, Basel
  - Site Reference ID/Investigator# 289, Geneva
  - Site Reference ID/Investigator# 243, Lausanne
  - Site Reference ID/Investigator# 254, Sankt Gallen
- Site Reference ID/Investigator# 241, Taipei, Taiwan
- United Kingdom (7):
  - Site Reference ID/Investigator# 238, Birmingham
  - Site Reference ID/Investigator# 232, Brighton
  - Site Reference ID/Investigator# 226, London
  - Site Reference ID/Investigator# 231, London
  - Site Reference ID/Investigator# 227, London
  - Site Reference ID/Investigator# 228, London
  - Site Reference ID/Investigator# 229, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 131 sites in 19 countries.
Pre-assignment Details: Of the 672 subjects randomized, 8 discontinued from the study prior to receiving study drug due to withdrawal of consent (3), acute illness (2), lost to follow-up (1), other (1), and required prohibited medication (1).
Groups:
- LPV/r 800/200 mg QD Tablet: lopinavir/ritonavir 800/200 mg once daily (QD) tablet
- LPV/r 800/200 mg QD SGC (Through Week 8): lopinavir/ritonavir 800/200 mg once daily (QD) soft gel capsule (SGC)
- LPV/r 400/100 mg BID Tablet: lopinavir/ritonavir 400/100 mg twice daily (BID) tablet
- LPV/r 400/100 mg BID SGC (Through Week 8): lopinavir/ritonavir 400/100 mg twice daily (BID) soft gel capsule (SGC)
Period: Study Start Through 8 Weeks
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8)
Started | 167 | 166 | 166 | 165
Completed | 163 | 161 | 155 | 160
Not Completed | 4 | 5 | 11 | 5
Not completed — Adverse Event | 1 | 2 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0
Not completed — Lost to Follow-up | 1 | 2 | 3 | 2
Not completed — Noncompliance | 0 | 0 | 2 | 2
Not completed — Death | 1 | 0 | 0 | 0
Period: Study Start Through 48 Weeks
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8)
Started | 333 (Number of subjects who started the study, not the number who completed the first 8 weeks.) | 0 (After Week 8, these subjects received the tablet formulation once daily through the end of study.) | 331 (Number of subjects who started the study, not the number who completed the first 8 weeks.) | 0 (After Week 8, these subjects received the tablet formulation twice daily through the end of study.)
Completed | 284 | 0 | 276 | 0
Not Completed | 49 | 0 | 55 | 0
Not completed — Adverse Event | 16 | 0 | 10 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 11 | 0
Not completed — Lost to Follow-up | 8 | 0 | 14 | 0
Not completed — Noncompliance | 3 | 0 | 8 | 0
Not completed — Death | 2 | 0 | 1 | 0
Not completed — Virologic failure | 2 | 0 | 4 | 0
Not completed — Relocated, Needed to take twice daily | 8 | 0 | 7 | 0
Period: Study Start Through 96 Weeks
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8)
Started | 333 (Number of subjects who started the study, not the number who completed the first 48 weeks.) | 0 (After Week 8, these subjects received the tablet formulation once daily through the end of study.) | 331 (Number of subjects who started the study, not the number who completed the first 48 weeks.) | 0 (After Week 8, these subjects received the tablet formulation twice daily through the end of study.)
Completed | 256 | 0 | 254 | 0
Not Completed | 77 | 0 | 77 | 0
Not completed — Adverse Event | 20 | 0 | 16 | 0
Not completed — Withdrawal by Subject | 15 | 0 | 13 | 0
Not completed — Lost to Follow-up | 19 | 0 | 18 | 0
Not completed — Noncompliance | 6 | 0 | 11 | 0
Not completed — Death | 2 | 0 | 2 | 0
Not completed — Virologic failure | 5 | 0 | 8 | 0
Not completed — Relocated, Needed to take twice daily | 10 | 0 | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8) | Total
Number analyzed (Participants) | 167 | 166 | 166 | 165 | 664
Age Continuous [Mean (Standard Deviation); unit: years] | 38.7 (9.80) | 38.2 (9.63) | 38.3 (9.69) | 39.5 (10.31) | 38.7 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 31 | 39 | 38 | 144
  Male | 131 | 135 | 127 | 127 | 520
CD4+ T Cell Count [Mean (Standard Deviation); unit: cells/mm3] — For once daily (QD) soft gel capsule (SGC), N=165.
  cells/mm3 | 209.9 (125.10) | 222.6 (127.37) | 226.4 (136.64) | 202.9 (139.57) | 215.5 (132.34)
Plasma HIV-1 RNA Level [Mean (Standard Deviation); unit: log10 copies/mL] | 4.92 (0.64) | 4.94 (0.67) | 5.04 (0.68) | 5.06 (0.64) | 4.99 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Adverse Events of Diarrhea During the First 8 Weeks
Time Frame: Week 8
Population: All randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Subjects
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8)
Number analyzed (Participants) | 167 | 166 | 166 | 165
Percentage of Subjects | 49.1 | 54.8 | 44.6 | 49.7
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 800/200 mg QD SGC (Through Week 8) vs LPV/r 400/100 mg BID Tablet vs LPV/r 400/100 mg BID SGC (Through Week 8); Cochran-Mantel-Haenszel (CMH) test stratified by dosing regimen was used to assess the null hypothesis of no difference between the tablet and soft gel capsule (SGC). Sample size was 600 subjects (150 each in the 4 groups). Based on a projected 48% reporting treatment-emergent diarrhea in the QD arm and 32% in the BID arm within the SGC group, with a 12% reduction in the corresponding tablet groups, this sample size provided 80% power to determine a difference between the tablet and SGC; Test type: Superiority or Other; p > 0.100, Cochran-Mantel-Haenszel

2. Primary Outcome: Percentage of Subjects With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Levels < 50 Copies/mL at Week 48
Time Frame: Week 48
Population: Intent-to-treat noncompleters considered failures (ITT, NC=F); all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Subjects
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8)
Number analyzed (Participants) | 333 | 0 | 331 | 0
Percentage of Subjects | 77.2 |  | 75.8 |
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 400/100 mg BID Tablet; The null hypothesis was that the response rate for the once daily (QD) regimen was more than 12% lower than the response rate for the twice daily (BID) regimen. The planned sample size of 600 subjects (300 subjects in each of the QD and BID treatment regimens) provided over 90% power to reject the null hypothesis, i.e., to determine noninferiority based on the 12% margin; Test type: Non-Inferiority or Equivalence — The 95% confidence interval for the difference in response rates (QD minus BID, based on the normal approximation to the binomial distribution) was used to assess noninferiority. The QD regimen was considered noninferior to the BID regimen if the lower limit of the confidence interval remained above -12%; p = 0.715, normal approx. to the binomial distr; percentage of subjects responding = 1.3, 95% CI [-5.1 to 7.8]

3. Secondary Outcome: Percentage of Subjects With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Levels < 50 Copies/mL at Week 96
Time Frame: Week 96 (End of Study)
Population: as for outcome 2
Measure: Number; unit: Percentage of Subjects
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8)
Number analyzed (Participants) | 333 | 0 | 331 | 0
Percentage of Subjects | 64.9 |  | 69.2 |
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 400/100 mg BID Tablet; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.249, normal approx. to the binomial distr; percentage of subjects responding = -4.3, 95% CI [-11.5 to 2.8]

4. Secondary Outcome: Mean Change From Baseline to Week 96 in CD4+ T Cell Counts
Time Frame: Week 96 (End of Study)
Population: All randomized subjects who received at least 1 dose of study drug and who had CD4+ T cell counts available at both the Baseline Visit and Week 96.
Measure: Mean (Standard Error); unit: cells/microliter
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 800/200 mg QD SGC (Through Week 8) | LPV/r 400/100 mg BID Tablet | LPV/r 400/100 mg BID SGC (Through Week 8)
Number analyzed (Participants) | 333 | 0 | 331 | 0
cells/microliter | 238.4 (10.02) |  | 254.0 (10.00) |
Statistical Analysis 1: Comparison: LPV/r 800/200 mg QD Tablet vs LPV/r 400/100 mg BID Tablet; Test type: Superiority or Other; p = 0.269, ANOVA

ADVERSE EVENTS:
Arm/Group | LPV/r 800/200 mg QD Tablet | LPV/r 400/100 mg BID Tablet
Serious Adverse Events (participants affected / at risk) | 37/333 | 50/331
Other Adverse Events (participants affected / at risk) | 292/333 | 287/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r 800/200 mg QD Tablet (N=333) | LPV/r 400/100 mg BID Tablet (N=331)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Lymphatic disorder (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Death (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 6
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Immune reconstitution syndrome (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Anogenital warts (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Meningitis tuberculous (Infections and infestations) | 1 | 0
Perichondritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 1 | 2
Typhoid fever (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood urine present (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Reversible ischemic neurological deficit (Nervous system disorders) | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Depression (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Drug dependence (Psychiatric disorders) | 1 | 0
Panic attack (Nervous system disorders) | 0 | 1
Psychotic disorder (Nervous system disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiform (Skin and subcutaneous tissue disorders) | 1 | 0
Granuloma skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Idiopathic capillaritis (Skin and subcutaneous tissue disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 2 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r 800/200 mg QD Tablet (N=333) | LPV/r 400/100 mg BID Tablet (N=331)
Abdominal pain (Gastrointestinal disorders) | 26 | 28
Abdominal pain upper (Gastrointestinal disorders) | 22 | 16
Diarrhea (Gastrointestinal disorders) | 210 | 197
Dyspepsia (Gastrointestinal disorders) | 21 | 9
Flatulence (Gastrointestinal disorders) | 17 | 27
Nausea (Gastrointestinal disorders) | 105 | 84
Vomiting (Gastrointestinal disorders) | 46 | 46
Asthenia (General disorders) | 25 | 18
Fatigue (General disorders) | 45 | 37
Influenza like illness (General disorders) | 9 | 19
Pyrexia (General disorders) | 28 | 29
Bronchitis (Infections and infestations) | 29 | 26
Gastroenteritis (Infections and infestations) | 9 | 19
Influenza (Infections and infestations) | 28 | 24
Nasopharyngitis (Infections and infestations) | 58 | 61
Sinusitis (Infections and infestations) | 19 | 17
Upper respiratory tract infection (Infections and infestations) | 29 | 25
Hypercholesterolemia (Metabolism and nutrition disorders) | 18 | 19
Hypertriglyceridemia (Metabolism and nutrition disorders) | 18 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 15
Dizziness (Nervous system disorders) | 16 | 17
Headache (Nervous system disorders) | 44 | 33
Anxiety (Psychiatric disorders) | 13 | 18
Depression (Psychiatric disorders) | 18 | 19
Insomnia (Psychiatric disorders) | 24 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 36
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 14
Rash (Skin and subcutaneous tissue disorders) | 27 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Provide ABBOTT at least thirty (30) days prior to submission for review, ABBOTT shall return comments within thirty (30) days of receipt of draft. Proposed draft shall be delayed an additional sixty (60) days in addition to the Review Period